CLINICAL TRIAL: NCT06352307
Title: Risk Stratification, Early Prevention and Treatment Strategies for Arrhythmogenic Cardiomyopathy (STARTER): a Multicenter Retro-prospective Cohort Study
Brief Title: Risk Stratification, Early Prevention and Treatment Strategies for Arrhythmogenic Cardiomyopathy
Acronym: STARTER
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-532
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Arrhythmogenic Cardiomyopathy
Keywords: Arrhythmogenic cardiomyopathy; Prognostic factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — For the retrospectively enrolled patients, we will collect their biological samples previously housed in the Biobank of The First Affiliated Hospital of Xi'an Jiaotong University.
  For the prospectively enrolled patients, we will collect a variety of biological samples at admission, before discharge, 1st, 3rd, 6th, 9th month, 1st, 2nd, 3rd year after discharge, including blood, urine, feces, other types of body fluids (such as pericardial effusion), tissue samples from surgery and biopsy (such as pericardial effusion, myocardial tissue, tumors, blood clots, etc.), or samples that need to be disposed of as medical waste (blood clots, etc.), or the sample itself requires pathological examination to assist in diagnosis and treatment (e.g. endocardial muscle biopsy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Right ventricular ACM group: The patients mainly had right ventricular enlargement and right ventricular fibrous adipose tissue replacement, and were diagnosed with right ventricular ACM.
  Interventions: Other: Diagnosis of ACM
- Left ventricular ACM group: The patients mainly had left ventricular enlargement and left ventricular fibroadipose tissue replacement, and were diagnosed with left ventricular ACM.
  Interventions: Other: Diagnosis of ACM
- Biventricular ACM group: The patients mainly had biventricular enlargement and fibroadipose tissue replacement, and were diagnosed with biventricular ventricular ACM.
  Interventions: Other: Diagnosis of ACM

INTERVENTIONS:
Other: Diagnosis of ACM — Definite ACM diagnosis is based on the consensus-based 2010 Task Force Criteria, which include major and minor criteria in six categories (depolarization and repolarization abnormalities, arrhythmia, imaging, histology, and family history/genetics). Among these, repolarization abnormalities (T-wave inversion in the precordial leads) constitute the most commonly observed, followed by frequent premature ventricular complex. With regards to imaging techniques, both the presence of wall motion abnormalities and an abnormal ventricular volume or function are required for fulfilment. Definite ACM consists of two major criteria or one major and two minor criteria or four minor criteria from different categories. Borderline ACM consists of one major and one minor criterion or three minor criteria from different categories.

SUMMARY:
This study will include patients diagnosed with Arrhythmogenic cardiomyopathy (ACM) in the First Affiliated Hospital of Xi 'an Jiaotong University and other centers, and collect clinical data and biological samples of patients with different ACM phenotypes. Through the establishment of disease cohort and long-term follow-up, to explore the disease characteristics, development law, clinical characteristics, natural course of disease and long-term prognosis of ACM.

DETAILED DESCRIPTION:
This study will include patients diagnosed with Arrhythmogenic cardiomyopathy (ACM) in the First Affiliated Hospital of Xi 'an Jiaotong University and other centers, and collect clinical data and biological samples of patients with different ACM phenotypes. Through the establishment of disease cohort and long-term follow-up, to explore the disease characteristics, development law, clinical characteristics, natural course of disease and long-term prognosis of ACM.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old.
* The diagnosis of ACM was confirmed by cardiac ultrasound, electrocardiogram, magnetic resonance angiography, pathological examination and gene sequencing.
* Patients or their families agreed to participate in the study and authorized informed consent.

Exclusion Criteria:

* Incomplete clinical data.
* Do not agree to the inclusion or refuse to authorize the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with ACM at all centers including The First Affiliated Hospital of Xi'an Jiaotong University.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2032-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in the incidence of mortality rate | At diagnosis, before discharge (about 7 days), 1, 3, 6, 9 month, 1, 2, 3 year.
  The survival status will be obtained from the medical records and phone calls to patients or their family members.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yan, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiantong University, Xi'an, Shaanxi, China